CLINICAL TRIAL: NCT02753348
Title: Copenhagen Baby Heart
Status: Completed | Type: Observational
Sponsor: Henning Bundgaard (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other); Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Sponsor-Investigator, Henning Bundgaard, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-16001518
Record Dates: First submitted 2016-04-24; First posted 2016-04-27 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample from umbilical cord for DNA extraction and analysis of biomarkers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newborns: Newborns (within 14 days from birth)
  Interventions: Other: Echocardiography; Other: Blood analysis from umbilical cord blood; Other: ECG; Other: Measurement of oxygen saturation

INTERVENTIONS:
Other: Echocardiography
Other: Blood analysis from umbilical cord blood
Other: ECG
Other: Measurement of oxygen saturation

SUMMARY:
Copenhagen Baby Heart is an observational, cohort study of >30.000 children born in the Copenhagen area 2016-2018.

Newborns are examined with echocardiography, electrocardiogram, measurements of oxygen saturation and analyses of umbilical cord blood.

The main objectives of the baseline assessments in Copenhagen Baby Heart are to assess the prevalence of congenital and inherited heart disease unrecognized prenatally, to assess the yield of routine echocardiography shortly after birth and to establish reference values for echocardiography in Danish neonates.

Prospective follow-up of the birth cohort is planned with the purpose to assess the life-long development of cardiovascular disease as well as other conditions and to study associations between both pre- and postnatal exposure and disease, including life style, environmental and genetic factors.

DETAILED DESCRIPTION:
Copenhagen Baby Heart is an observational, cohort study of >30.000 children born in the Copenhagen area 2016-2018.

Purpose

* To assess the prevalence of congenital and inherited heart disease not detected prenatally, e.g. bicuspid aortic valve.
* To assess the diagnostic and clinical yield of routine echocardiography in neonates.
* To establish reference values for echocardiography and ECG for Danish neonates.
* To establish reference values for routine biochemical analyses in umbilical cord blood.
* To assess the prevalence of familial hypercholesterolemia in Danish newborns.
* To assess the life-long development of cardiovascular disease as well as other conditions and to study associations between both pre- and postnatal exposure and disease, including life style, environmental and genetic factors.

Methods Approximately 18.000 children are born yearly in the Copenhagen area. From 1. April 2016 - 1. April 2018 the parents of all newborns will be offered enrollment in the research project when attending a routine prenatal ultrasound.

Investigators plan to enroll >30.000 newborns.

After birth, blood is drawn from the umbilical chord and immediately analyzed for routine biochemical markers. Samples will also be stored for future biochemical analyses and DNA sequencing.

Within the first 14 days of life the children are examined with standardized echocardiography, electrocardiogram and measurements of oxygen saturation.

Information about maternal and paternal health including inherited disorders within the family as well as information about the pregnancy and birth are collected in a central database.

Follow-up When indicated children will be followed clinically. For research-purposes, prospective, register-based follow-up is planned for the entire birth cohort and with clinical visits for sub-groups of the population.

ELIGIBILITY:
Inclusion Criteria:

* Born at one of three hospitals in the Copenhagen area

Exclusion Criteria:

* Failure of providing consent (parents)

Ages: 0 Weeks to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns (0-14 days old, or for preterms when >2000g) born at three different hospitals in the Copenhagen area.
Sampling Method: Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2016-04; Primary Completion 2018-10 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of congenital heart defects | 2 years

REFERENCES:
- [Derived] Farooqui AF, Norsk JB, Raja AA, Hjortdal V, Bjerrekaer JK, Fagerlund MR, Vogg RO, Pihl C, Bundgaard H, Iversen K, Sillesen AS. Prevalence of Congenital Aortic Valve Regurgitation in a Newborn Cohort. Pediatr Cardiol. 2026 Jan 20. doi: 10.1007/s00246-025-04149-0. Online ahead of print. PMID 41555067
- [Derived] Sillesen AS, Jorgensen FS, Petersen OB, Zingenberg H, Dannesbo S, Raja AA, Vogg ROB, Vejlstrup N, Iversen K, Bundgaard H. Difference in pre- and postnatal prevalence of congenital cardiac tumors in a large population-based cohort. Acta Obstet Gynecol Scand. 2025 Oct;104(10):1875-1882. doi: 10.1111/aogs.70018. Epub 2025 Aug 5. PMID 40763039
- [Derived] Blixenkrone-Moller E, Dannesbo S, Dehn AM, Pihl CA, Sillesen AS, Vogg ROB, Raja AA, Colan S, Mertens L, Vejlstrup N, Bundgaard H, Iversen K. Interatrial Communications: Prevalence and Subtypes in 12,385 Newborns-a Copenhagen Baby Heart Study. Pediatr Cardiol. 2025 Aug;46(6):1570-1580. doi: 10.1007/s00246-024-03571-0. Epub 2024 Jul 13. PMID 39003423
- [Derived] Molin J, Hartmann J, Paerregaard MM, Thygesen CB, Sillesen AS, Raja AA, Vogg ROB, Iversen KK, Bundgaard H, Christensen AH. The Neonatal QRS Complex and Its Association with Left Ventricular Mass. Pediatr Cardiol. 2024 Feb;45(2):248-256. doi: 10.1007/s00246-023-03361-0. Epub 2023 Dec 27. PMID 38151605
- [Derived] Norregaard MMO, Basit S, Sillesen AS, Raja AA, Jorgensen FS, Iversen KK, Bundgaard H, Boyd HA, Vogg ROB. Impact of maternal age and body mass index on the structure and function of the heart in newborns: a Copenhagen Baby Heart Study. BMC Med. 2023 Dec 18;21(1):499. doi: 10.1186/s12916-023-03207-9. PMID 38110921
- [Derived] Dehn AM, Paerregaard MM, Sellmer A, Dannesbo S, Blixenkrone-Moller E, Sillesen AS, Raja AA, Iversen KK, Bundgaard H, Christensen AH, Hjortdal V. Electrocardiographic Characteristics in 438 Neonates with Atrial Septal Defects. Pediatr Cardiol. 2024 Mar;45(3):580-587. doi: 10.1007/s00246-023-03324-5. Epub 2023 Nov 1. PMID 37914855
- [Derived] Paerregaard MM, Hartmann J, Sillesen AS, Pihl C, Dannesbo S, Kock TO, Pietersen A, Raja AA, Iversen KK, Bundgaard H, Christensen AH. The Wolff-Parkinson-White pattern in neonates: results from a large population-based cohort study. Europace. 2023 Jul 4;25(7):euad165. doi: 10.1093/europace/euad165. PMID 37465966
- [Derived] Dehn AM, Dannesbo S, Sellmer A, Hoffner L, Blixenkrone-Moller E, Sillesen AS, Raja AA, Vejlstrup N, Iversen K, Bundgaard H, Hjortdal V. Atrial Septal Defect: Larger Right Ventricular Dimensions and Atrial Volumes as Early as in the First Month After Birth-a Case-Control Study Including 716 Neonates. Pediatr Cardiol. 2023 Oct;44(7):1578-1586. doi: 10.1007/s00246-023-03211-z. Epub 2023 Jun 27. PMID 37369832
- [Derived] Paerregaard MM, Hartmann J, Vogg O, Pietersen A, Boyd HA, Raja AA, Iversen KK, Bundgaard H, Christensen AH. The Impact of Maternal Age on the Neonatal Electrocardiogram. Neonatology. 2022;119(5):629-637. doi: 10.1159/000524439. Epub 2022 Jul 20. PMID 35858538
- [Derived] Borresen MF, Blixenkrone-Moller E, Kock TO, Sillesen AS, Vogg ROB, Pihl CA, Norsk JB, Vejlstrup NG, Christensen AH, Iversen KK, Bundgaard H, Axelsson Raja A. Prevalence of Left Ventricular Noncompaction in Newborns. Circ Cardiovasc Imaging. 2022 Jun;15(6):e014159. doi: 10.1161/CIRCIMAGING.121.014159. Epub 2022 Jun 21. PMID 35727876
- [Derived] Hartmann J, Paerregaard MM, Norsk J, Pietersen A, Iversen KK, Bundgaard H, Christensen AH. Gestational Age and Neonatal Electrocardiograms. Pediatrics. 2021 Dec 1;148(6):e2021050942. doi: 10.1542/peds.2021-050942. PMID 34814190
- [Derived] Paerregaard MM, Kock J, Pihl C, Pietersen A, Iversen KK, Bundgaard H, Christensen AH. The Evolution of the Neonatal QRS Axis during the First Four Weeks of Life. Neonatology. 2021;118(2):155-162. doi: 10.1159/000513526. Epub 2021 Mar 10. PMID 33691309
- [Derived] Sillesen AS, Pihl C, Raja AA, Davidsen AS, Lind LE, Dannesbo S, Navne J, Raja R, Vejlstrup N, Lange T, Bundgaard H, Iversen K. Repeatability and Reproducibility of Neonatal Echocardiography: The Copenhagen Baby Heart Study. J Am Soc Echocardiogr. 2019 Jul;32(7):895-905.e2. doi: 10.1016/j.echo.2019.02.015. Epub 2019 May 7. PMID 31076139
- [Derived] Sillesen AS, Raja AA, Pihl C, Vogg ROB, Hedegaard M, Emmersen P, Sundberg K, Tabor A, Vedel C, Zingenberg H, Kruse C, Wilken-Jensen C, Nielsen TH, Jorgensen FS, Jeppesen DL, Sondergaard L, Kamstrup PR, Nordestgaard BG, Frikke-Schmidt R, Vejlstrup N, Boyd HA, Bundgaard H, Iversen K. Copenhagen Baby Heart Study: a population study of newborns with prenatal inclusion. Eur J Epidemiol. 2019 Jan;34(1):79-90. doi: 10.1007/s10654-018-0448-y. Epub 2018 Oct 10. PMID 30306423